CLINICAL TRIAL: NCT04654390
Title: A Multi-center, Randomized, Double-Blind, Active-controlled, Phase3, Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of DWP16001 in Patients With Type 2 Diabetes Mellitus
Brief Title: The Efficacy Nad Safety of DWP16001 Compared to Active Drug in the Treatment of Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP16001303
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP16001 Amg, Dapagiflozin Bmg placebo (Experimental): Tablets, Orally, Once daily
  Interventions: Drug: DWP16001 Amg
- DWP16001 Amg placebo, Dapagliflozin Bmg (Active Comparator): Tablets, Orally, Once daily
  Interventions: Drug: DWP16001 Amg

INTERVENTIONS:
Drug: DWP16001 Amg — Tablets, Orally, Once daily

SUMMARY:
The purpose of this study is to determine the efficacy and safety of DWP16001 compared to active drug in the treatment of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 80 years
2. Subjects with 7% ≤ HbA1c ≤ 11% at Screening
3. Subjects with BMI of 20-45 kg/m2

Exclusion Criteria:

1. Different type of diabetes mellitus which is not T2DM (type 1 diabetes mellitus, secondary diabetes mellitus, or congenital renal glucosuria)
2. Symptoms of stress urinary incontinence, dysuria that is not controlled by medications due to neurogenic bladder or prostatic hyperplasia, anuria, oliguria, or urinary retention
3. Severe diabetes complications (proliferative diabetic retinopathy, nephropathy of stage 4 or higher, or serious diabetic neuropathy)
4. eGFR < 60 mL/min/1.73 m2
5. Severe gastrointestinal diseases: active ulcer, gastrointestinal or rectal bleeding, active inflammatory bowel syndrome, biliary duct obstruction, active gastritis that is not controlled by medication, etc.
6. Uncontrolled hypertension (SBP >180 mmHg or DBP > 110 mmHg)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Change from Visit 2(Randomization) in HbA1c level at Week 24 after administation of the IP | at Week 24
  HbA1c level at Week 24 after administration of the IP

SECONDARY OUTCOMES:
Changes from Visit 2 (randomization) in HbA1c level at Weeks 6, 12, and 18 after administration of the IP | at weeks 6, 12, and 18
  HbA1c level at Weeks 6, 12, and 18 after administration of the IP
Changes from Visit 2 (randomization) in FPG level at Weeks 6, 12, 18, and 24 after administration of the IP | at weeks 6, 12, 18, and 24
  FPG level at Weeks 6, 12, 18, and 24 after administration of the IP
Proportions of subjects who achieved HbA1c level < 7% at Weeks 6, 12, 18, and 24 after administration of the IP | at weeks 6, 12, 18, and 24
  HbA1c level < 7% at Weeks 6, 12, 18, and 24 after administration of the IP

CONTACTS AND LOCATIONS:
Overall Officials: Sungrae KIm, MD, PhD, Study Director — The Catholic University of Korea Bucheon St. Mary's Hospital, Republic of Korea
Locations (1):
- The Catholic University of Korea Bucheon St. Mary's Hospital, Republic of Korea, Bucheon-si, South Korea

IPD SHARING:
Plan to Share IPD: No